CLINICAL TRIAL: NCT01540903
Title: Controlled Human Malaria Infection by Intradermal Injection of Plasmodium Falciparum Sporozoites (PfSPZ Challenge)in Tanzanian Adults
Brief Title: Controlled Human Malaria Infection by Intradermal Injection of Plasmodium Falciparum Sporozoites in Tanzanian Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sanaria Inc. (Industry)
Collaborators: Ifakara Health Research and Development Centre (Other); Swiss Tropical & Public Health Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: BSPZC1
Record Dates: First submitted 2012-02-23; First posted 2012-02-29 (Estimated); Last update posted 2014-09-10 (Estimated); Status verified 2014-09

CONDITIONS: Malaria
Keywords: Malaria Challenge; Plasmodium falciparum; PfSPZ Challenge; Controlled; human; malaria infection
MeSH Terms: conditions — Malaria; Malaria, Falciparum | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Group 1 10,000 PfSPZ (Experimental): 12 volunteers, ID PfSPZ Challenge total dose 10,000 PfSPZ administered by 2 injections of 50µL each.
  Interventions: Biological: PfSPZ Challenge
- Group 2 25,000 PfSPZ (Experimental): 12 volunteers, ID PfSPZ Challenge total dose 25,000 PfSPZ administered in 4 injections of 10µL each.
  Interventions: Biological: PfSPZ Challenge
- Controls - saline (Placebo Comparator): 4 Volunteers, ID saline administered in 2 injections of 50µL each and 2 volunteers, ID saline administered in 4 injections of 10µL each.
  Interventions: Biological: Saline

INTERVENTIONS:
Biological: PfSPZ Challenge — Aseptic, purified, vialed, cryopreserved, fully infectious NF54 Plasmodium falciparum sporozoites (PfSPZ Challenge)
  Other Names: Plasmodium falciparum sporozoites
  Arms: Group 1 10,000 PfSPZ; Group 2 25,000 PfSPZ
Biological: Saline — Saline
  Arms: Controls - saline

SUMMARY:
The proposed trial will evaluate whether relatively non immune populations in endemic countries can be effectively infected with aseptic, purified, cryopreserved sporozoites (PfSPZ Challenge) given intradermally.

DETAILED DESCRIPTION:
Controlled human malaria infection (CHMI) is a critical component of malaria vaccine and drug development and is an important element of any strategy for accelerating the development of new tools for malaria control, elimination and eradication. Until now, CHMI has been performed in malaria naïve subjects from countries not endemic for malaria using both infectious mosquitoes and recently, aseptic, purified, cryopreserved Plasmodium falciparum sporozoites (PfSPZ). Results from these studies report significant infection success in all study subjects and an excellent safety profile.

The conduct of CHMI studies in malaria endemic populations will allow early understanding of responses to new vaccines and drugs in endemic country populations and for direct comparisons between previously exposed and non-exposed individuals. Performing CHMI studies in malaria endemic countries will reduce associated costs, speed-up the process of testing and substantially contribute to the acceleration of the malaria vaccine and drug research and development processes.

This study to be conducted in Bagamoyo, Tanzania, aims to see whether people in endemic countries with minimal previous history of malaria are suitable for CHMI using PfSPZ Challenge. This study will also assess whether the success rate of the experiment is improved by lowering the volume of injection and increasing the number of inoculations. Hence, the study will contribute towards improvements in the CHMI studies using syringe and needle inoculation of sporozoites.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Male aged between 20-35 years, healthy volunteers
* Good Health status based on history & clinical examination
* Residing in or near DaresSalaam
* Willing to contribute to science in Tanzania
* Free from malaria parasite by blood smear & qRT-PCR
* Not suffering from any chronic illness including HIV/AIDS
* No documented history of malaria infection for the past 5 yrs
* Able & willing to come for complete one year follow up including minimum of three weeks of hospitalization
* All volunteers must sign the informed consent form & answer correctly 15 out 15 questions demonstrating their understanding of the meaning & procedures of the study
* Volunteer agrees to inform study doctor & agrees to release medical information concerning contra-indications for participation in the study
* Living with a third party that will contact the study team if in case of alteration of consciousness during the first month of the study
* Willing to undergo a Pf sporozoite challenge.
* Willing to take curative treatment for malaria (Coartem®) & any other medication which may be prescribed by a study doctor during study period
* All volunteers agree to stay in the hospital during parts of the study (overnight after challenge, up to 15 days during follow up & 3 days of Coartem® treatment)
* Reachable (24/7) by mobile phone during the whole study period
* Agreement not to participate in another study during the study period.
* Agreement not to donate blood during the study period.
* Available to attend all study visits
* Willingness to undergo HIV, hepatitis B & hepatitis C tests

Exclusion Criteria:

* History of malaria in the past 5 yrs
* Plans to travel outside the Dar-es-salaam or Coast Region in first month (day 0-28) of the study
* Plans to travel to highly malarious areas in the 6 months following the study period
* Previous participation in malaria vaccine study &/or positive serology for Plasmodium falciparum asexual crude extract antibodies above acceptable cut off established for the site.
* History of arrhythmias or prolonged QT-interval or other cardiac disease
* Positive family history of in the 1st & 2nd degree relative for cardiac disease <50 yrs old.
* Volunteers unable to read & write in English & give written informed consent
* Previous history of drug or alcohol abuse interfering with normal social function
* A history of psychiatric disease
* The use of chronic immunosuppressive drugs, antibiotics, or other immune modifying drugs within three months of study onset (inhaled & topical corticosteroids are allowed) & during the study period
* A history or confirmed sickle cell anemia, sickle cell trait, thalassemia , thalassemia trait or G6PD deficiency
* Co-worker of the Ifakara Health Institute
* Symptoms, physical signs & laboratory values suggestive of systemic disorders including renal, hepatic, cardiovascular, pulmonary, skin, immunodeficiency, psychiatric, & other conditions which could interfere with the interpretation of the study results or compromise the health of the volunteers
* History of diabetes mellitus or cancer
* An estimated, ten year risk of fatal cardiovascular disease of <5%, as estimated by the Systematic Coronary Risk Evaluation (SCORE) system
* Clinically significant abnormalities in electrocardiogram at screening
* Body Mass Index below 18 or above 30kg/m2
* Any clinically significant deviation from the normal range in biochemistry or hematology blood tests or in urine analysis or electrolytes
* Positive HIV, Hepatitis B virus or Hepatitis C Virus tests
* Participation in any other clinical study within 30 days prior to the onset of the study or during the study period
* Volunteers unable to be closely followed for social, geographic or psychological reasons
* Known hypersensitivity of other contra-indications to Coaterm® or Malarone® including treatment taken by the volunteer that interferes with Coartem® or Malarone®
* Any confirmed or suspected immunosuppressive or immunodeficient condition, including asplenia

Ages: 20 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2012-02; Primary Completion 2012-09 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Number of volunteers positive in each group through day 28 of follow up. | 5 to 28 days
  Thick smears will be performed according to a standard operating procedure. In short, 15 μL of whole blood will be distributed on standardized 3-well slides, providing an equal slide thickness for all smears. Slides are dried and stained with Giemsa. 200 fields per slide will be read at 1000X. Slides are considered positive if they contain 2 or more parasites per 200 fields.

SECONDARY OUTCOMES:
Time from inoculation until first positive parasitemia by thick smear in each volunteer in the two groups. | 5-28 days
Time from inoculation to until first positive parasitemia by qRT-PCR in each volunteer in the two groups. | 5-28 days
  qRT-PCR will be performed according to standard procedure described in Hermsen et al. Mol. Biochem. Parasitol. 2001; 118: 247-251. In short, qRT-PCR will be performed on the multicopy 18S ribosomal RNA gene. Cultured P. falciparum ring stage parasites are taken as a positive control. All samples are spiked with murine white blood cells, and a murine albumin gene PCR is used to determine efficacy of DNA isolation.
Kinetics of parasitemia in positive volunteers in the two groups as measured by qRT-PCR. | 5-28 days
  Thick smear, malaria rapid diagnostic test and qRT-PCR samples will be taken from the same 3 mL EDTA vacutainer tube. Histidine Rich Protein 2 based malaria rapid diagnostic tests will be used in parallel to thick smears.
Occurrence or intensity of signs or symptoms in the two groups of volunteers | 5 days to 6 months
  Signs and symptoms will be recorded at all visits and whenever a trial volunteer reports signs or symptoms to the trial physician between visits. The following signs and symptoms will be solicited: fever, headache, malaise, fatigue, myalgia, arthralgia, nausea, vomiting, chills, diarrhea, abdominal pain (Verhage, Telgt, Bousema, Hermsen, van Gemert, van der Meer, & Sauerwein 2005), chest pain, palpitations and shortness of breath.

CONTACTS AND LOCATIONS:
Overall Officials: Salim Abdulla, MD, PhD, Principal Investigator — Ifakara Health Institute (IHI), Tanzania
Locations (1):
- Bagamoyo Research and Training Center, Ifakara Health Institute, Bagamoyo, Tanzania

REFERENCES:
- [Result] Shekalaghe S, Rutaihwa M, Billingsley PF, Chemba M, Daubenberger CA, James ER, Mpina M, Ali Juma O, Schindler T, Huber E, Gunasekera A, Manoj A, Simon B, Saverino E, Church LWP, Hermsen CC, Sauerwein RW, Plowe C, Venkatesan M, Sasi P, Lweno O, Mutani P, Hamad A, Mohammed A, Urassa A, Mzee T, Padilla D, Ruben A, Sim BKL, Tanner M, Abdulla S, Hoffman SL. Controlled human malaria infection of Tanzanians by intradermal injection of aseptic, purified, cryopreserved Plasmodium falciparum sporozoites. Am J Trop Med Hyg. 2014 Sep;91(3):471-480. doi: 10.4269/ajtmh.14-0119. Epub 2014 Jul 28. PMID 25070995